CLINICAL TRIAL: NCT01970878
Title: A 28-Week, Multi-Center, Randomized, Double Blind, Parallel-Group, Active-Controlled Safety Extension Study to Evaluate the Safety and Efficacy of PT003, PT001, and PT005 in Subjects With Moderate to Very Severe COPD, With Spiriva® Handihaler® as an Active Control
Brief Title: Extension Study to Evaluate the Safety and Efficacy of PT003, PT001, and PT005 in Subjects With Moderate to Very Severe COPD, With Spiriva® Handihaler® (PINNACLE 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT003008-00
Record Dates: First submitted 2013-10-18; First posted 2013-10-28 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GFF MDI (PT003) (Experimental)
  Interventions: Drug: GFF MDI (PT 003)
- GP MDI (PT001) (Experimental)
  Interventions: Drug: GP MDI (PT001)
- FF MDI (PT005) (Experimental)
  Interventions: Drug: FF MDI (PT005)
- Open-label tiotropium bromide inhalation powder (Active Comparator): Open-label tiotropium bromide inhalation powder (Spiriva® Handihaler®)
  Interventions: Drug: Open-label tiotropium bromide inhalation (Spiriva® Handihaler®)

INTERVENTIONS:
Drug: GFF MDI (PT 003) — GFF MDI administered as two puffs BID
  Arms: GFF MDI (PT003)
Drug: GP MDI (PT001) — GP MDI administered as two puffs BID
  Arms: GP MDI (PT001)
Drug: FF MDI (PT005) — FF MDI administered as two puffs BID
  Arms: FF MDI (PT005)
Drug: Open-label tiotropium bromide inhalation (Spiriva® Handihaler®) — Taken as 1 capsule daily containing 18 μg of open-label tiotropium via the Handihaler dry powder inhaler (DPI)
  Arms: Open-label tiotropium bromide inhalation powder

SUMMARY:
This is a multi-center, randomized, double-blind, parallel group, chronic dosing, active-controlled, 28-week safety extension study of the two pivotal 24-week safety and efficacy studies (Studies PT003006 and PT003007). This study is designed to assess the long-term safety and tolerability of Glycopyrrolate (GP) and Formoterol Fumarate (FF) combination (GFF) metered dose inhaler (MDI), GP MDI, and FF MDI in subjects with moderate to very severe COPD over a total observation period of 52 weeks. Open-label Spiriva is included as an active control. To be eligible for this study, a subject must complete participation in Study PT003006 (NCT01854645) or Study PT003007 (NCT01854658).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant in/completion of previous 24-week PINNACLE Phase III Trial.
* Male or female subjects at least 40 years of age and no older than 80 at Visit 1.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* Subjects with FEV1/forced vital capacity (FVC) ratio of <0.70 and FEV1 <80% predicted normal and ≥750 mL if FEV1 <30% of predicted normal value.
* Subjects willing and, in the opinion of the investigator, able to adjust current COPD therapy as required by the protocol

Key Exclusion Criteria:

* Significant diseases other than COPD, i.e. disease or condition which, in the opinion of the investigator, may put the patient at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study
* Current diagnosis of asthma or alpha-1 antitrypsin deficiency
* Other active pulmonary disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or uncontrolled sleep apnea
* Hospitalized due to poorly controlled COPD within 3 months prior to screening or during the Screening Period
* Poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to screening or during the Screening Period
* Lower respiratory tract infections that required antibiotics within 6 weeks prior to screening or during the Screening Period
* Unstable ischemic heart disease, left ventricular failure, or documented myocardial infarction within 12 months of enrollment.
* Recent history of acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft within the past three months
* Congestive heart failure (CHF) New York Heart Association (NYHA) Class III/IV)
* Clinically significant abnormal 12-lead electrocardiogram (ECG)
* Abnormal liver function tests defined as alanine transaminase (ALT), aspartate transaminanse (AST), or total bilirubin ≥ 1.5 times upper limit of normal at Visit 1 and on repeat testing
* Cancer not in complete remission for at least five years
* History of hypersensitivity to β2-agonists, glycopyrronium or other muscarinic anticholinergics, lactose/milk protein or any component of the MDI

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Chair — Pearl Therapeutics, Inc.
Locations (125):
- United States (110):
  - Pearl Investigative Site, Andalusia, Alabama
  - Pearl Investigative Site, Anniston, Alabama
  - Pearl Investigative Site, Athens, Alabama
  - Pearl Investigative Site, Birmingham, Alabama
  - Pearl Investigative Site, Jasper, Alabama
  - Pearl Investigative Site, Glendale, Arizona
  - Pearl Investigative Site, Mesa, Arizona
  - Pearl Investigative Site, Phoenix, Arizona
  - Pearl Investigative Site, Scottsdale, Arizona
  - Pearl Investigative Site, Tucson, Arizona
  - Pearl Investigative Site, Anaheim, California
  - Pearl Investigative Site, Carlsbad, California
  - Pearl Investigative Site, Lakewood, California
  - Pearl Investigative Site, Los Angeles, California
  - Pearl Investigative Site, Monterey Park, California
  - Pearl Investigative Site, Pasadena, California
  - Pearl Investigative Site, Poway, California
  - Pearl Investigative Site, Sacramento, California
  - Pearl Investigative Site, San Diego, California
  - Pearl Investigative Site, Tustin, California
  - Pearl Investigative Site, Vista, California
  - Pearl Investigative Site, Colorado Springs, Colorado
  - Pearl Investigative Site, Denver, Colorado
  - Pearl Investigative Site, Fort Collins, Colorado
  - Pearl Investigative Site, Wheat Ridge, Colorado
  - Pearl Investigative Site, Danbury, Connecticut
  - Pearl Investigative Site, Waterbury, Connecticut
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Miami, Florida
  - Pearl Investigative Site, Ormond Beach, Florida
  - Pearl Investigative Site, Panama City, Florida
  - Pearl Investigative Site, Pensacola, Florida
  - Pearl Investigative Site, St. Petersburg, Florida
  - Pearl Investigative Site, Tampa, Florida
  - Pearl Investigative Site, Winter Park, Florida
  - Pearl Investigative Site, Atlanta, Georgia
  - Pearl Investigative Site, Austell, Georgia
  - Pearl Investigative Site, Columbus, Georgia
  - Pearl Investigative Site, Duluth, Georgia
  - Pearl Investigative Site, Gainesville, Georgia
  - Pearl Investigative Site, Couer D'aline, Idaho
  - Pearl Investigative Site, Champaign, Illinois
  - Pearl Investigative Site, Evanston, Illinois
  - Pearl Investigative Site, Peoria, Illinois
  - Pearl Investigative Site, River Forest, Illinois
  - Pearl Investigative Site, Avon, Indiana
  - Pearl Investigative Site, Evansville, Indiana
  - Pearl Investigative Site, South Bend, Indiana
  - Pearl Investigative Site, Iowa City, Iowa
  - Pearl Investigative Site, Olathe, Kansas
  - Pearl Investigative Site, Topeka, Kansas
  - Pearl Investigative Site, Louisville, Kentucky
  - Pearl Investigative Site, Lafayette, Louisiana
  - Pearl Investigative Site, Sunset, Louisiana
  - Pearl Investigative Site, Hollywood, Maryland
  - Pearl Investigative Site, Livonia, Michigan
  - Pearl Investigative Site, Southfield, Michigan
  - Pearl Investigative Site, Edina, Minnesota
  - Pearl Investigative Site, Fridley, Minnesota
  - Pearl Investigative Site, Minneapolis, Minnesota
  - Pearl Investigative Site, Woodbury, Minnesota
  - Pearl Investigative Site, Chesterfield, Missouri
  - Pearl Investigative Site, Springfield, Missouri
  - Pearl Investigative Site, St Louis, Missouri
  - Pearl Investigative Site, Bellvue, Nebraska
  - Pearl Investigative Site, Omaha, Nebraska
  - Pearl Investigative Site, Las Vegas, Nevada
  - Pearl Investigative Site, Albuquerque, New Mexico
  - Pearl Investigative Site, Corning, New York
  - Pearl Investigative Site, Burlington, North Carolina
  - Pearl Investigative Site, Charlotte, North Carolina
  - Pearl Investigative Site, Greensboro, North Carolina
  - Pearl Investigative Site, Huntersville, North Carolina
  - Pearl Investigative Site, Mooresville, North Carolina
  - Pearl Investigative Site, Raleigh, North Carolina
  - Pearl Investigative Site, Wilmington, North Carolina
  - Pearl Investigative Site, Winston-Salem, North Carolina
  - Pearl Investigative Site, Cincinnati, Ohio
  - Pearl Investigative Site, Dayton, Ohio
  - Pearl Investigative Site, Bend, Oregon
  - Pearl Investigative Site, Brandon, Oregon
  - Pearl Investigative Site, Medford, Oregon
  - Pearl Investigative Site, Portland, Oregon
  - Pearl Investigative Site, Philadelphia, Pennsylvania
  - Pearl Investigative Site, Pittsburgh, Pennsylvania
  - Pearl Investigative Site, Charleston, South Carolina
  - Pearl Investigative Site, Easley, South Carolina
  - Pearl Investigative Site, Gaffney, South Carolina
  - Pearl Investigative Site, Murrells Inlet, South Carolina
  - Pearl Investigative Site, Rock Hill, South Carolina
  - Pearl Investigative Site, Spartanburg, South Carolina
  - Pearl Investigative Site, Rapid City, South Dakota
  - Pearl Investigative Site, Bristol, Tennessee
  - Pearl Investigative Site, Johnson City, Tennessee
  - Pearl Investigative Site, Kingsport, Tennessee
  - Pearl Investigative Site, Austin, Texas
  - Pearl Investigative Site, Houston, Texas
  - Pearl Investigative Site, Huntsville, Texas
  - Pearl Investigative Site, Longview, Texas
  - Pearl Investigative Site, New Braunfels, Texas
  - Pearl Investigative Site, San Antonio, Texas
  - Pearl Investigative Site, Midvale, Utah
  - Pearl Investigative Site, Salt Lake City, Utah
  - Pearl Investigative Site, South Burlington, Vermont
  - Pearl Investigative Site, Abingdon, Virginia
  - Pearl Investigative Site, Richmond, Virginia
  - Pearl Investigative Site, Spokane, Washington
  - Pearl Investigative Site, Tacoma, Washington
  - Pearl Investigative Site, Morgantown, West Virginia
  - Pearl Investigative Site, West Allis, Wisconsin
- Australia (9):
  - Pearl Investigative Site, New Lambton, New South Wales
  - Pearl Investigative Site, Westmead, New South Wales
  - Pearl Investigative Site, Brisbane, Queensland
  - Pearl Investigative Site, Cairns, Queensland
  - Pearl Investigative Site, Wooloongabba, Queensland
  - Pearl Investigative Site, Adelaide, South Australia
  - Pearl Investigative Site, Heidelberg, Victoria
  - Pearl Investigative Site, Nederlands, Western Australia
  - Pearl Investigative Site, Perth, Western Australia
- New Zealand (6):
  - Pearl Investigative Site, Otahuhu, Aukland
  - Pearl Investigative Site, Caversham, Dunedin
  - Pearl Investigative Site, Greenlabe, East Aukland
  - Pearl Investigative Site, Hamilton, Waikato Region
  - Pearl Investigative Site, Newtown, Wellington Region
  - Pearl Investigative Site, Tauranga

REFERENCES:
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 205 sites from November 2013- December 2014. The entire study period was a maximum of 30 weeks.
Pre-assignment Details: Study PT003008 was an extension of Studies NCT01854645 and NCT01854658. A proportion of subjects on active treatment were randomly invited to participate. Analysis of Study PT003008 included all subjects enrolled in the lead-in studies to avoid bias. Hence, the number analyzed will be greater than the 892 subjects enrolled into the extension.
Groups:
- GFF MDI (PT003): GFF MDI 14.4/9.6 mcg
- GP MDI (PT001): GP MDI 14.4 mcg
- FF MDI (PT005): FF MDI 9.6 mcg
- Spiriva® Handihaler® (Open-label): Open-label tiotropium bromide inhalation powder 18 mcg
Period: Overall Study
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label)
Started | 290 | 218 (218 subjects were reported in the CSR, 1 had no completion status) | 213 | 171
Completed | 253 | 191 | 187 | 147
Not Completed | 37 | 27 | 26 | 24
Not completed — Withdrawal by Subject | 11 | 10 | 14 | 7
Not completed — Lost to Follow-up | 1 | 3 | 2 | 4
Not completed — Administrative Reasons | 1 | 0 | 0 | 4
Not completed — Lack of Efficacy | 2 | 1 | 2 | 0
Not completed — Adverse Event | 12 | 7 | 4 | 3
Not completed — Protocol Specified Criteria | 10 | 4 | 3 | 6
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — No Completion Status | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population includes all subjects enrolled into active treatment arms for the lead-in Studies PT003006 & PT003007
Groups:
- Total: Total of all reporting groups
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Total
Number analyzed (Participants) | 1035 | 888 | 884 | 450 | 3257
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.3) | 62.8 (8.4) | 62.8 (8.1) | 62.9 (8.6) | 62.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 473 | 392 | 392 | 182 | 1439
  Male | 562 | 496 | 492 | 268 | 1818

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning -Pre-dose Trough FEV1 Over 52 Weeks
Description: Change From Baseline in Morning Pre-Dose Trough FEV1 Over 52 Weeks as a Model-Based Average (ITT Population). FEV1 was assessed at multiple time points post-baseline, and a model-based average of all visits starting from Week 2 through week 52 inclusive was calculated. The change values reported in the table represent the change between the baseline and the average FEV1 post-baseline.
Time Frame: Baseline and Weeks 2 to 52
Population: Subjects in the ITT population from the lead-in studies who had data for the parameter.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label)
Number analyzed (Participants) | 1021 | 872 | 871 | 445
Liters | 0.133 [0.122 to 0.144] | 0.076 [0.064 to 0.088] | 0.068 [0.056 to 0.080] | 0.107 [0.091 to 0.124]

2. Secondary Outcome: Self-Administered Computerized (SAC) TDI Focal Score Over 52 Weeks
Description: SAC TDI focal score over 52 Weeks as a Model-Based Average (ITT Population) The TDI is an instrument which measures the changes in the participant's dyspnea from Baseline. The scores in the TDI evaluate ratings for 3 different categories (functional impairment, magnitude of task in exertional capacity, and magnitude of effort). TDI scores ranged from -3 (major deterioration) to +3 (major improvement); total score = -9 to 9.
Time Frame: Baseline and Weeks 4 to 52
Population: Subjects in the ITT population from the lead-in studies who had data for the parameter.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label)
Number analyzed (Participants) | 1002 | 867 | 871 | 442
Scores on a scale | 0.5 [0.4 to 0.6] | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.4] | 0.4 [0.3 to 0.6]

3. Secondary Outcome: Peak Change From Baseline in FEV1 Within 2 Hrs Post-dosing
Description: Peak change from Baseline FEV1 Over 52 Weeks is a Model-Based Average (ITT Population). Peak FEV1 was assessed at multiple visits post-baseline, and a model-based average of all visits starting from Week 2 through week 52 inclusive was calculated. The change values reported in the table represent the change between the baseline and the average Peak FEV1 post-baseline.
Time Frame: Baseline and Weeks 2 to 52
Population: Subjects in the ITT population from the lead-in studies who had data for the parameter.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label)
Number analyzed (Participants) | 1035 | 888 | 883 | 450
Liters | 0.363 [0.351 to 0.375] | 0.234 [0.221 to 0.247] | 0.275 [0.262 to 0.288] | 0.270 [0.251 to 0.288]

4. Secondary Outcome: Change From Baseline in SGRQ Total Score
Description: The SGRQ is a disease-specific questionnaire, self-completed by participants, used to evaluate the effect of GFF MDI, FF MDI and GP MDI on health-related quality of life as compared to placebo in subjects with COPD. The scores range from 0 (best possible health status) to 100 (worst possible health status). The SGRQ contains 76 items grouped into three domains (symptoms, activity and impacts). Change from Baseline in total score of -4 units or lower is considered as clinically meaningful improvement in quality of life. SGRQ Total Score was assessed at multiple visits post-baseline, and a model-based average of all visits starting from Week 12 through week 52 inclusive was calculated. The change values reported in the table represent the change between the baseline and the average SGRQ Total Score post-baseline.
Time Frame: Baseline and Weeks 12 to 52
Population: Subjects in the ITT population from the lead-in studies who had data for the parameter
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label)
Number analyzed (Participants) | 995 | 843 | 845 | 434
Scores on a scale | -3.3 [-4.0 to -2.6] | -1.9 [-2.7 to -1.2] | -2.4 [-3.2 to -1.7] | -2.9 [-4.0 to -1.8]

5. Secondary Outcome: Change From Baseline in Average Daily Rescue Ventolin Use
Description: Subjects recorded in their diary the number of puffs of rescue Ventolin HFA taken on each study day. The subject's average daily number of puffs of rescue Ventolin HFA was calculated over the entire 52-week treatment period. Missing values were ignored in both the numerator and denominator. Diary data recorded during the last 7 days of the 10-14 day screening period were used to calculate the baseline average. Change in rescue Ventolin HFA use was calculated by subtracting the baseline average from the 52-week average.
Time Frame: Baseline through Week 52
Population: Subjects in the ITT population from the lead-in studies who had data for the parameter
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs per day
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label)
Number analyzed (Participants) | 1035 | 885 | 881 | 447
Puffs per day | -0.9 [-1.0 to -0.7] | -0.4 [-0.6 to -0.3] | -0.7 [-0.8 to -0.5] | -0.4 [-0.6 to -0.1]

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: The Safety Population was similar to the ITT Population (all subjects who were randomized to active [non-placebo] treatment in Study PT003006 or Study PT003007 and received at least 1 dose of the study treatment in Study PT003006 or Study PT003007, regardless of whether or not they participated in Study PT003008).
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label)
Serious Adverse Events (participants affected / at risk) | 114/1036 | 90/890 | 78/890 | 49/451
Other Adverse Events (participants affected / at risk) | 109/1036 | 77/890 | 90/890 | 51/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (PT003) (N=1036) | GP MDI (PT001) (N=890) | FF MDI (PT005) (N=890) | Spiriva® Handihaler® (Open-label) (N=451)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 32 (32) | 30 (33) | 19 (19) | 12 (12)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 15 (15) | 14 (14) | 4 (4) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical Pneuomonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis Staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extradural Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Opthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Operative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urospepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiglottic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocelluar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 4 (4) | 2 (3) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (4)
Acute myocardial infrarction (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atriventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio myopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occulsion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial iscaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Upper gastrointestinal haemmorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestial haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large Intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 4 (4) | 3 (3) | 4 (4) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (PT003) (N=1036) | GP MDI (PT001) (N=890) | FF MDI (PT005) (N=890) | Spiriva® Handihaler® (Open-label) (N=451)
Nasopharyngitis (Infections and infestations) | 70 (74) | 38 (40) | 55 (61) | 28 (28)
Upper Respiratory Tract Infection (Infections and infestations) | 39 (42) | 39 (44) | 35 (38) | 23 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.